CLINICAL TRIAL: NCT06293313
Title: The Effect of Mindfulness Practice on Coping With Primary Dysmenorrhea on Pain and Anxiety Level
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Simge Ozturk, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Inonu-SBF-SO-03
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Dysmenorrhea; Anxiety; Anxiety Disorders and Symptoms; Pain, Menstrual
Keywords: mindfulness; pain; anxiety; dysmenorrhea; nursing
MeSH Terms: conditions — Dysmenorrhea; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: A total of two groups, a control group and a experimental group wo mindfulness group
Who Masked: Investigator, Outcomes Assessor
Masking Description: The determination of which university would be included in the control and experimental groups in the research was made through a randomization method. The selection was done blindly by an independent academician unrelated to the research. As a result of the randomization, the control group and the experimental groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness group (Experimental): Students who agree to participate in the research will be met with students in a quiet room of the school by making an appointment. Individuals will be pre-tested. Mindfulness will be applied within the first 3 days of the menstrual period. After continuing the training for 8 weeks, an interim test will be applied. After 3 months, the final test will be applied
  Interventions: Procedure: Mindfulness training
- Control Group (Sham Comparator): Students in the control group will not be given any application. A pre-test will be administered before starting the study, an interim test will be applied 8 weeks after the pre-test, and a post-test will be applied 3 months after the interim test. After the study is over, mindfulness will be applied to the students in the control group.
  Interventions: Other: Will not be given any application

INTERVENTIONS:
Procedure: Mindfulness training — Before starting the study, an appointment will be made to meet with the students participating in the mindfulness group with randomization on the specified day and time. The students and the researcher will meet in a quiet, calm room of the school. Students will be informed about the practice of mindfulness and their written and verbal consents will be obtained before participating in the study. Then, a pre-test will be applied to the students who agree to participate in the study.
  Arms: Mindfulness group
Other: Will not be given any application — Before starting the research, the students in the control group determined by the randomization method will be informed about the research. Written and verbal consent will be obtained from the students that the students agree to participate in the research. Afterwards, students will meet in a quiet and calm room of the school on the specified day and time. Before starting the research, students will be given a pre-test. A mid-term test will be performed 8 weeks after the pre-test.
  Arms: Control Group

SUMMARY:
The aim of this project is to determine the effect of mindfulness practice to cope with dysmenorrhea on pain and anxiety levels. The project will be carried out in a semi-randomized controlled manner. It will be applied to 100 students with dysmenorrhea (100 students by increasing by 10%, taking into account the losses that may occur in the 90 students determined in the sample calculation). Students who meet the inclusion criteria and approve of participating in the project will be given a pre-test before the application. 'Introductory Information Form', 'VAS Scale' and 'State and Trait Anxiety Scale' will be used in the pre-test. After the pre-test, mindfulness practice will be applied for 8 weeks (1 day/120 minutes per week). At the end of 8 weeks, an intermediate test will be performed in the first 3 days of the first menstrual cycle. After the mid-term test, students will practice mindfulness on their own with the brochures provided. Motivational messages will be sent to students for mindfulness practice, starting 3 days before their cycle. The final test will be administered 3 months after the intermediate test. 'VAS Scale' and 'State and Trait Anxiety Scale' will be used in the mid-test and post-test.

DETAILED DESCRIPTION:
Dysmenorrhea is a gynecological condition that negatively affects the lives of more than half of women during menstruation. The severity of dysmenorrhea can be mild, moderate or high. Dysmenorrhea negatively affects women's social relations, daily lives, business lives, academic achievements and quality of life. Pharmacological and non-pharmacological treatments are used in its treatment. Among the non-pharmacological methods used in the treatment of dysmenorrhea, methods such as aromatherapy, yoga, massage, regular exercise, acupuncture, acupressure, TENS and cognitive behavioral therapy have been used. Mindfulness, one of the cognitive behavioral treatment methods, reduces stress, anxiety and depression in women. The aim of this project is to determine the effect of mindfulness practice to cope with dysmenorrhea on pain and anxiety levels. The project will be carried out in a semi-randomized controlled manner. It will be applied to 100 students with dysmenorrhea (100 students by increasing by 10%, taking into account the losses that may occur in the 90 students determined in the sample calculation). Students who meet the inclusion criteria and approve of participating in the project will be given a pre-test before the application. 'Introductory Information Form', 'VAS Scale' and 'State and Trait Anxiety Scale' will be used in the pre-test. After the pre-test, mindfulness practice will be applied for 8 weeks (1 day/120 minutes per week). At the end of 8 weeks, an intermediate test will be performed in the first 3 days of the first menstrual cycle. After the mid-term test, students will practice mindfulness on their own with the brochures provided. Motivational messages will be sent to students for mindfulness practice, starting 3 days before their cycle. The final test will be administered 3 months after the intermediate test. 'VAS Scale' and 'State and Trait Anxiety Scale' will be used in the mid-test and post-test.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Being literate,
* Having dysmenorrhea,
* Volunteering to participate in the study,
* Participating in mindfulness practice for 8 weeks,
* Not using any pharmacological or non-pharmacological methods,
* Studying at Bartin University

Exclusion Criteria:

* Not being a university student
* Not experiencing dysmenorrhea
* Not attending at least two mindfulness practices

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female students who are 18 years of age or older studying at the university will be included.
Enrollment: 200 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-08-28 (Estimated)

PRIMARY OUTCOMES:
VAS Pain Scale | five month
  The scale consists of a horizontal line of 100 mm in length. At the left end of the line is the phrase "No pain" or "The pain is completely gone", while at the right end is the phrase "Unbearable pain" or "No reduction in pain at all". The patient is instructed to mark a point on the line that will accurately reflect his or her own pain. The distance of the patient's sign to the left end is measured. This distance, usually measured in millimeters, is reported as "points".

SECONDARY OUTCOMES:
State and Trait Anxiety Scale | five month
  Anxiety Inventory includes two separate scales consisting of a total of forty items. There are ten reversed expressions in the State Anxiety Scale and these are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. In the Trait Anxiety Scale, there are seven reversed expressions and these are items 21, 26, 27, 30, 33, 36 and 39. The feelings or behaviors expressed in the State Anxiety Scale items are answered by marking one of the following options: (1) not at all, (2) a little, (3) a lot and (4) completely, according to the severity of such experiences. The emotions or behaviors expressed in the Trait Anxiety Scale are marked according to their frequency as (1) almost never, (2) sometimes, (3) most of the time and (4) almost always. The total score obtained from each scale varies between 20 and 80. A high score indicates a high level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Simge Öztürk, Ph.D, Principal Investigator — Bartın Unıversity
Locations (1):
- Bartin University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No